CLINICAL TRIAL: NCT01382901
Title: A Phase 2a Study Evaluating the Efficacy and Safety of a Novel Intravenous (IV) Iron Preparation (VIT-45) in the Treatment of Restless Legs Syndrome (RLS)
Brief Title: Intravenous (IV) Iron Preparation (VIT-45) in the Treatment of Restless Legs Syndrome (RLS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1VIT05009
Record Dates: First submitted 2011-02-23; First posted 2011-06-27 (Estimated); Results first posted 2011-06-27 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-01

CONDITIONS: Restless Legs Syndrome (RLS)
MeSH Terms: conditions — Restless Legs Syndrome | interventions — ferric carboxymaltose

ARMS (2):
- Intravenous (IV) Iron (Experimental)
  Interventions: Drug: Ferric Carboxymaltose (FCM)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ferric Carboxymaltose (FCM)
  Other Names: VIT-45
  Arms: Intravenous (IV) Iron
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the safety of 2 dosage regimens of Intravenous (IV) iron Ferric Carboxymaltose (FCM) in comparison to placebo in patients with Restless Legs Syndrome (RLS)

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects > or = to 18 years old, and able to give informed consent to the study.
* RLS signs and symptoms affirming diagnosis. The IRLS Diagnostic Criteria for RLS must be met.
* Subjects have RLS symptoms > or = to 5 nights per week for at least the past 3 months.
* A baseline score > or = to 15 on the IRLS Rating Scale.
* At least one leg with an average baseline Periodic Leg Movement while asleep (PLMS) > or = to 15 movements per hour and at least 3 days of baseline PLMS data is measurable in each leg.
* Subjects on anti-depressants, sleep medications, dopamine agonists, benzodiazepines, narcotics or other RLS treatments must be off therapy at least one week or 5 half lives, whichever is longer before any baseline RLS assessments and PLM measurements are obtained.
* Subject has regular sleep hours between 9 p.m. and 9 a.m.
* Subjects at risk for pregnancy must have a negative pregnancy test at baseline and be practicing an acceptable form of birth control.

Exclusion Criteria:

* RLS 2° to other CNS disease or injury. Such disorders include peripheral neuropathy, neurodegenerative disorders, and multiple sclerosis.
* RLS 2° to Chronic Kidney Disease.
* Any pain related or sleep related disorders (e.g. sleep apnea) which may confound the outcome measures.
* History of neuroleptic akathisia.
* Oral iron use (including multivitamins with iron) after screening.
* Parenteral iron use within 4 weeks prior to screening.
* Parenteral iron use > 125 mg per week within 4 to 8 weeks prior to screening.
* History of > or = to 10 blood transfusions in the past 2 years.
* Anticipated need for blood transfusion during the study.
* Known hypersensitivity reaction to any component to FCM.
* Previously participated in an FCM clinical trial.
* Chronic or serious active severe infection.
* Malignancy (other than basal or squamous cell skin cancer or the subject has been cancer free for > 5 years).
* Active inflammatory arthritis (e.g. rheumatoid arthritis, SLE).
* Receiving prescription medication for the treatment of bronchospasm.
* Pregnant or lactating women.
* Severe peripheral vascular disease with significant skin changes.
* Seizure disorder currently being treated with medication.
* Baseline ferritin > 300 ng/mL.
* Baseline TSAT > or = to 45%.
* History of hemochromatosis or hemosiderosis or other iron storage disorders.
* AST or ALT greater than the upper limit of normal.
* Hemoglobin greater than the upper limit of normal.
* Calcium or phosphorous outside the normal range.
* Known positive hepatitis B antigen (HBsAg) or hepatitis C viral antibody (HCV) with evidence of active hepatitis.
* Known positive HIV-1/HIV-2 antibodies (anti-HIV).
* Received an investigational drug within 30 days before randomization.
* Chronic alcohol or drug abuse within the past 6 months.
* Significant cardiovascular disease, including myocardial infarction within 12 months prior to study inclusion, congestive heart failure NYHA (New York Heart Association) III or IV, or poorly controlled hypertension according to the judgment of the investigator.
* Any other pre-existing laboratory abnormality, medical condition or disease which in view of the investigator participation in this study may put the subject at risk.
* Subject unable to comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-03; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Period: March 23, 2006 to July 16, 2007 Locations: Hospitals and Medical Clinics (15 total sites)
Groups:
- Ferric Carboxymaltose (FCM) 2 x 500 mg: 500mg intravenous (IV) dose of FCM on Day 0 and Day 5.
- Placebo: Intravenous (IV) solution of placebo on Day 0 and Day 5.
Period: Overall Study
Arm/Group | Ferric Carboxymaltose (FCM) 2 x 500 mg | Placebo
Started | 24 | 21
Completed | 7 | 7
Not Completed | 17 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ferric Carboxymaltose (FCM) 2 x 500 mg | Placebo | Total
Number analyzed (Participants) | 24 | 21 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 15 | 35
  >=65 years | 4 | 6 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (11.42) | 54.1 (13.68) | 51.7 (12.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 11 | 28
  Male | 7 | 10 | 17
Region of Enrollment [Number; unit: participants]
  United States | 24 | 21 | 45

OUTCOME MEASURES:

1. Primary Outcome: International Restless Legs Syndrome (IRLS) Total Score
Description: The scale represents the patients symptoms of RLS. The patient rates his/her symptoms based on 10 questions with a maximum possible score of 40 representing the most severe symptoms while a score of 0 represents no symptoms at all.
Time Frame: Change from Baseline to Day 28
Population: Evaluable Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ferric Carboxymaltose (FCM) 2 x 500 mg | Placebo
Number analyzed (Participants) | 24 | 19
Scores on a scale | -8.9 (8.52) | -4.0 (0.040)

ADVERSE EVENTS:
Time Frame: 1 year and 4 months
Arm/Group | Ferric Carboxymaltose (FCM) 2 x 500 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/21
Other Adverse Events (participants affected / at risk) | 9/24 | 6/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ferric Carboxymaltose (FCM) 2 x 500 mg (N=24) | Placebo (N=21)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Blood phosphorus decreased (Investigations) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less